CLINICAL TRIAL: NCT07167095
Title: Evaluation of Factors Affecting 90-Day Mortality After Emergency Department Discharge in Patients With Advanced Cancer
Brief Title: 90-Day Mortality After Emergency Department Discharge in Advanced Cancer
Acronym: CARE-90
Status: Completed | Type: Observational
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Galip Can Uyar, Medical Oncologist, Ankara Etlik City Hospital
Other Study IDs: AEŞH-BADEK2-2025-242; AEŞH-BADEK2-2025-242 (Other: Etlik City Hospital Scientific Research and Evaluation Ethics Committee)
Record Dates: First submitted 2025-08-24; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Advanced Cancer; Mortality; Oncology; Emergency Department Admission; Metastatic Solid Tumors
Keywords: 90-Day Mortality; Emergency Department; Prognostic Factors; Performance Status; Nutritional and Inflammatory Markers; Oncology Supportive Care; Palliative Care
MeSH Terms: conditions — Neoplasms; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Advanced Cancer Patients Presenting to the Emergency Department: This retrospective cohort includes adult patients (≥18 years) with pathologically confirmed stage IV solid tumors who presented to the emergency department of Etlik City Hospital between December 2022 and March 2025. Patients were eligible if they had received systemic anticancer therapy within the previous 6 months and had complete clinical and laboratory records. Both patients discharged from the ED and those who were admitted or died during the ED visit are included. Data collected include demographic characteristics, performance status, primary tumor type, metastatic sites, reasons for ED admission, laboratory values, and subsequent outcomes. The cohort will be analyzed to identify prognostic factors associated with 90-day mortality, ED re-admissions, and re-hospitalizations.
  Interventions: Other: Retrospective Data Collection and Analysis

INTERVENTIONS:
Other: Retrospective Data Collection and Analysis — This intervention refers to retrospective evaluation of clinical and laboratory data of advanced cancer patients who presented to the emergency department between December 2022 and March 2025. Data will be extracted from the hospital information system (HBYS) and national death registry (e-Nabız). Parameters include demographics, ECOG performance status, primary tumor type, metastatic sites, laboratory markers (e.g., NLR, CRP, albumin, LDH), and outcomes such as 90-day mortality, re-admissions, and re-hospitalizations. No experimental treatment, drug, or device is administered as part of the study.
  Other Names: Observational Chart Review

SUMMARY:
This retrospective observational study investigates factors associated with 90-day mortality among patients with advanced cancer who present to the emergency department (ED). The study will include stage IV solid tumor patients who visited the ED of Etlik City Hospital between December 2022 and March 2025. Demographic, clinical, and laboratory parameters such as performance status, nutritional and inflammatory markers, and biochemical values will be analyzed. The primary objective is to identify prognostic indicators that predict short-term mortality following ED visits. By establishing risk profiles, the study aims to optimize patient triage, guide timely referral to supportive and palliative care services, and improve overall care strategies for advanced cancer patients in acute settings.

DETAILED DESCRIPTION:
Patients with advanced-stage cancer frequently present to emergency departments (EDs) due to complications related to disease progression, treatment side effects, or acute clinical deterioration. Such unplanned visits represent a critical point in the trajectory of cancer care, as they are often associated with poor short-term outcomes, repeated hospitalizations, and increased healthcare burden. Identifying reliable predictors of mortality following ED discharge is therefore essential for improving triage processes, tailoring management strategies, and ensuring timely referral to supportive or palliative care.

This retrospective cohort study will evaluate prognostic factors associated with 90-day mortality among patients with stage IV solid tumors presenting to the ED of Etlik City Hospital between December 2022 and March 2025. The study population will consist of patients who were discharged on the same day, admitted to the hospital, or who died during their ED visit. Clinical data will be retrieved from the hospital information system, and mortality outcomes will be verified using both institutional records and the national death registry.

Collected parameters will include demographic variables (age, sex, body mass index, smoking history), disease characteristics (primary tumor type, metastatic sites, prior systemic treatment), performance status (ECOG score), and laboratory values routinely obtained during ED visits (hemoglobin, leukocyte and platelet counts, neutrophil-to-lymphocyte ratio, C-reactive protein, albumin, lactate dehydrogenase, renal and liver function tests, and electrolytes). The primary endpoint will be 90-day all-cause mortality after ED presentation. Secondary outcomes will include in-hospital mortality during ED stay, 30-day ED re-admission rates, and 90-day re-hospitalizations.

Statistical analyses will be conducted to assess associations between clinical and laboratory variables and short-term mortality. Group comparisons will be performed using chi-square tests, Fisher's exact test, independent t-test, or Mann-Whitney U test, as appropriate. Multivariable logistic regression models will identify independent predictors of 90-day mortality, while Kaplan-Meier and Cox regression analyses will explore survival differences across patient subgroups stratified by ECOG status, albumin, BMI, and inflammatory markers. Post-hoc power analysis will be conducted to ensure robustness of the findings.

Existing literature highlights the prognostic significance of poor performance status, malnutrition, and systemic inflammation in cancer patients presenting to EDs. Low serum albumin (<3.5 g/dL), high neutrophil-to-lymphocyte ratio, low hemoglobin, and elevated LDH have consistently been associated with higher mortality risk. Similarly, unplanned ED visits often correlate with advanced disease burden, impaired quality of life, and reduced survival. However, most available studies are limited by small sample sizes, heterogeneous populations, or lack of integration between clinical and laboratory data. By analyzing a large cohort of 1,250-1,650 patients from a single tertiary cancer center, this study aims to overcome these limitations and provide a more comprehensive understanding of risk profiles in this vulnerable population.

The findings are expected to contribute valuable insights into the early identification of high-risk patients at the time of ED admission. Ultimately, these results could support the development of evidence-based prognostic models that inform clinical decision-making, improve allocation of healthcare resources, and enhance the integration of supportive and palliative care interventions for patients with advanced malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Pathologically confirmed stage IV (metastatic) solid malignancy
* Followed at Etlik City Hospital, Department of Medical Oncology
* Presented to the emergency department between December 2022 and March 2025
* Either discharged on the same day, admitted to the hospital, or died during the ED visit
* Received systemic anticancer therapy (chemotherapy, immunotherapy, targeted therapy, or hormonal therapy) within the past 6 months
* Availability of complete clinical and laboratory data

Exclusion Criteria:

* Stage I-III cancer patients
* Patients not receiving systemic therapy, only palliative/supportive care
* Patients followed in other oncology centers but presenting to Etlik City Hospital ED
* Patients with hematologic malignancies (e.g., leukemia, lymphoma, multiple myeloma)
* Patients with missing clinical or laboratory data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients (aged 18 years and older) with stage IV solid tumors who presented to the emergency department of Etlik City Hospital (Ankara, Türkiye) between December 2022 and March 2025. Eligible patients must have received systemic anticancer therapy within the preceding 6 months. Both patients discharged from the ED and those who were hospitalized or who died during their ED visit are included. The estimated enrollment is 1,250 patients.
Sampling Method: Non-Probability Sample
Enrollment: 1250 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
90-Day All-Cause Mortality After Emergency Department Visit | 90 days after emergency department visit
  All-cause mortality within 90 days following presentation to the emergency department among patients with stage IV solid tumors. Mortality status will be confirmed using the hospital information system (HBYS) and the national death registry (e-Nabız). Both in-hospital and out-of-hospital deaths will be included.

SECONDARY OUTCOMES:
In-Hospital Mortality During Emergency Department Visit | 30 days after ED discharge
  Proportion of patients with stage IV solid tumors who die during the index emergency department visit. Mortality will be confirmed via hospital records.
30-Day Emergency Department Re-admission | 30 days after ED discharge
  Proportion of patients discharged from the emergency department who return within 30 days for any cause. Re-admissions will be verified through hospital records.
90-Day Hospital Re-admission Rate | 90 days after ED discharge
  Proportion of patients discharged from the ED who are subsequently hospitalized within 90 days. Re-hospitalizations will be tracked using the hospital information system.
Correlation between ECOG Performance Status and 90-Day Mortality | 90 days after ED visit
  Eastern Cooperative Oncology Group (ECOG) Performance Status scale, which ranges from 0 (fully active) to 4 (completely disabled)
Correlation between Body Mass Index (BMI) and 90-Day Mortality | 90 days after ED visit
  BMI (kg/m²), calculated from body weight (kg) and height (m²) recorded in hospital records.
Correlation between CRP/Albumin Ratio and 90-Day Mortality | 90 days after ED visit
  CRP/Albumin ratio (mg/L ÷ g/dL), derived from laboratory test results in hospital records
Correlation between Neutrophil-to-Lymphocyte Ratio (NLR) and 90-Day Mortality | 90 days after ED visit
  Neutrophil-to-Lymphocyte Ratio, calculated from absolute neutrophil and lymphocyte counts in hospital laboratory records
Correlation between Hemoglobin and 90-Day Mortality | 90 days after ED visit
  Hemoglobin concentration (g/dL), measured by standard hospital laboratory tests
Correlation between Lactate Dehydrogenase (LDH) and 90-Day Mortality | 90 days after ED visit
  Lactate Dehydrogenase (U/L), measured by standard hospital laboratory tests

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No